CLINICAL TRIAL: NCT03309709
Title: Efficacy of Subcutaneous Progesterone in Premenopausal Woman With Endometrial Polyp: a Multicentric Randomized Control Trial
Brief Title: Endometrial Polyps Regression With Progesterone Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Roberta Venturella, Principal investigator, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Progesterone Polyps
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Endometrial Polyp

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- watch-and-wait patients (No Intervention): patients who receive a watch-and-wait approach
- Progesterone patients (Experimental): Treatment consists of 7 days of 25 mg subcutaneous progesterone administered from 18° to 25° day of the menstrual cycle and repeated for 3 cycles
  Interventions: Drug: subcutaneous progesterone

INTERVENTIONS:
Drug: subcutaneous progesterone — 25mg daily for 7 days
  Other Names: Pleyris
  Arms: Progesterone patients

SUMMARY:
This prospective randomized study will compare the regression rates of women managed with watch-and-wait approach and of those treated with 3 cycles of luteal 25mg subcutaneous progesterone from 18 to 25 days of menstrual cycle

DETAILED DESCRIPTION:
In premenopause, 25% of endometrial polyps regresses spontaneously in 1 year. According to guidelines, given that most premenopausal polyps are not malignant, there is an option for expectant approach with no surgical intervention. Studies on the efficacy of medical treatments for endometrial polyps are also recommended by gynaecologic societies, with the aim of finding cost-saving not invasive strategies to manage this common pathology. Up to now, nobody has investigated the effect of progestin administration on polyps, but molecular and clinical data suggest that the antiestrogenic effect of this hormone can be exploited to increase and speed-up their regression rate. Our preliminary results on the effect of three months of progesterone demonstrated a regression rate of 47,5% in women treated vs 12,5% in those don't receiving treatment.

Accordingly, in this prospective randomized study we aim to compare the regression rates of women managed with watch-and-wait approach and of those treated with 3 cycles of luteal 25mg subcutaneous progesterone from 18 to 25 days of menstrual cycle

ELIGIBILITY:
Inclusion Criteria:

* ultrasound diagnosis of endometrial polyps no more than 30 days before the enrollment
* signed informed consent

Exclusion Criteria:

* estrogenic and\or progestinic therapy two months before the enrollment
* tamoxifen therapy
* pelvic inflammatory disease
* gynaecologic neoplasia
* previous chemotherapy and radiotherapy
* autoimmune diseases, chronic disease, metabolic, and endocrine (hyperandrogenism, hyperprolactinemia, diabetes mellitus and thyroid disease)
* menopause
* Hypogonadotropic hypogonadism
* drugs causing menstrual irregularities

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-10-08 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Polyps regression rate | three months after the starting of treatment or of watch-wait approach
  US evidence of normal endometrial line without evidence of polyps

SECONDARY OUTCOMES:
Polyps dimensions | three months after the starting of treatment or of watch-wait approach
  Effect of progesterone on polyps dimensions measured in mm
Correlation between polyps dimension and regression | three months after the starting of treatment or of watch-wait approach
  Correlation between the size of the polyps and the efficacy of progesterone therapy in terms of regression of lesions
Side effects | three months after the starting of treatment
  Evaluation of any side effects
Progesterone effects on menstrual bleeding assessed with PBAC (Pictorial blood loss assesment chart) score | three months after the starting of treatment
  Effect of progestogen therapy on symptoms possibly present in patients with endometrial polyps, assessed with PBAC (Pictorial blood loss assesment chart) score.
  Patients will be asked to fill in the PBAC score during the first menstrual period following diagnosis and during the three months of medical treatment or watch and wait approach. The "8-days PBAC score" is an objective method used to quantify menstrual blood loss; according to this method, each patient records the extent of uterine bleeding during the first 8 days of menstrual cycle, quantizing it in terms of daily change in diapers and number/size of the clots. Each option has a numeric value (1=no bleeding; 2=spotting; 3=1-8 diapers per day; 4=heavy bleeding) and, based on the result obtained, the monthly PBAC score varies from 0 (amenorrhea) to > 500 (heavy bleeding). Menorrhagia occurs when PBAC score is >100 during a menstrual cycle, corresponding to a blood loss greater than 80 ml.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Venturella, MD, Principal Investigator — Magna Graecia University of Catanzaro
Locations (2):
- Italy (2):
  - Ospedale Pugliese Ciaccio, Catanzaro, Calabria
  - Federico II University, Naples

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venturella R, Miele G, Cefali K, Lico D, D'Alessandro P, Arduino B, Di Cello A, Zullo F, Di Carlo C. Subcutaneous Progesterone for Endometrial Polyps in Premenopausal Women: A Preliminary Retrospective Analysis. J Minim Invasive Gynecol. 2019 Jan;26(1):143-147. doi: 10.1016/j.jmig.2018.04.023. Epub 2018 May 2. PMID 29729409